CLINICAL TRIAL: NCT02046980
Title: Treatment of Apogeotropic Horizontal Canal Benign Paroxysmal Positional Vertigo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, HyunAh Kim, Assistant Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DK-0001
Record Dates: First submitted 2014-01-25; First posted 2014-01-28 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo | interventions — Vibration; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gufoni (Experimental): Gufoni maneuver for apogeotropic horizontal BPPV at the first day
  Interventions: Procedure: Gufoni
- Vibration (Experimental): Vibration maneuver for apogeotropic horizontal BPPV at the first day
  Interventions: Procedure: Vibration
- Sham (Sham Comparator): Sham maneuver for apogeotropic horizontal BPPV at the first day
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Gufoni
  Arms: Gufoni
Procedure: Vibration
  Arms: Vibration
Procedure: Sham
  Arms: Sham

SUMMARY:
To determine the short term therapeutic efficacies of Gufoni maneuver and mastoid oscillation in apogeotropic type of benign paroxysmal positional vertigo (BPPV) involving the horizontal semicircular canal (HC-BPPV), a randomized, prospective, sham-controlled study was conducted.

DETAILED DESCRIPTION:
The apogeotropic type of benign paroxysmal positional vertigo involving the horizontal canal (HC-BPPV) is likely due to otolithic debris in the anterior arm of the canal (canalithiasis) or the debris attached to the cupula (cupulolithiasis). It is important to seek the method to convert treatment-resistant apogeotropic form to the more treatment-responsive geotropic form in HC-BPPV. Recent randomized trials demonstrated that head shaking maneuver was more effective than the modified Semont maneuver and the Gufoni and head shaking maneuvers showed similar efficacy in treating apogeotropic HC-BPPV. Moreover, new repositioning maneuver using mastoid vibration showed good efficacies in patients with apogeotropic HC-BPPV in recent study. So we tried to compare the short term therapeutic efficacies of Gufoni maneuver and mastoid oscillation in apogeotropic HC-BPPV with a randomized, prospective, sham-controlled study.

ELIGIBILITY:
Inclusion Criteria:

1. history of vertigo associated with changes in head position
2. direction-changing horizontal nystagmus beating toward the uppermost ear (apogeotropic nystagmus) in both turning positions detected with Frenzel glasses or videoculography in the Head turning test
3. vertigo associated with the elicited nystagmus
4. symptom within 2 weeks
5. put one's signature on consent

Exclusion Criteria:

1. patients with identifiable central nervous system disorders that could explain the positional vertigo and nystagmus
2. the patients with apogeotropic form which was transited from geotropic after previous therapeutic maneuvers
3. the patients who transited from apogeotropic from vertical canal BPPV during study
4. patients who had possible cause of secondary BPPV such as Meniere's disease, migraine or recent trauma history
5. patients whose affected ear cannot be identified
6. patients with multiple canal atypical positional nystagmus or who were treated previously with repositioning maneuvers were excluded.
7. patients with cervical or lumbar spine problem

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Ah Kim, Study Director — Daegu KyungBook Dizziness society; Hyung Lee, Study Chair — Keimyung University Dongsan Medical Centerl
Locations (1):
- Daegu Kyungbook Dizziness society, Daegu, South Korea

REFERENCES:
- [Derived] Kim HA, Park SW, Kim J, Kang BG, Lee J, Han BI, Seok JI, Chung EJ, Kim J, Lee H. Efficacy of mastoid oscillation and the Gufoni maneuver for treating apogeotropic horizontal benign positional vertigo: a randomized controlled study. J Neurol. 2017 May;264(5):848-855. doi: 10.1007/s00415-017-8422-2. Epub 2017 Feb 20. PMID 28220291

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 217 patients enrolled in the study but 8 retracted their agreements.
Groups:
- Gufoni: Gufoni maneuver for apogeotropic horizontal benign paroxysmal positional vertigo (BPPV) at the first day
  Gufoni
- Vibration: Vibration maneuver for apogeotropic horizontal BPPV at the first day
  Vibration
- Sham: Sham maneuver for apogeotropic horizontal BPPV at the first day
  Sham
Period: Overall Study
Arm/Group | Gufoni | Vibration | Sham
Started | 72 | 72 | 73
Completed | 70 | 67 | 72
Not Completed | 2 | 5 | 1

BASELINE CHARACTERISTICS:
Population: 217 patients enrolled in the study but 8 retracted their agreements.
Groups:
- Gufoni: Gufoni maneuver for apogeotropic horizontal BPPV at the first day
  Gufoni
- Total: Total of all reporting groups
Arm/Group | Gufoni | Vibration | Sham | Total
Number analyzed (Participants) | 70 | 67 | 72 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.00 (11.58) | 62.22 (13.25) | 61.44 (13.48) | 61.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 39 | 52 | 133
  Male | 28 | 28 | 20 | 76
Symptom duration [Mean (Full Range); unit: days] | 3.37 [0 to 14] | 2.70 [0 to 14] | 2.52 [0 to 14] | 2.9 [0 to 14]
Lesion side [Number; unit: participants]
  Right side | 41 | 37 | 33 | 111
  Left side | 29 | 30 | 39 | 98

OUTCOME MEASURES:

1. Primary Outcome: Conversion in Direction of Nystagmus From Apogeotropic to Geotropic or Disappearance of Nystagmus
Time Frame: 2 days
Population: 217 patients enrolled in the study but 8 retracted their agreements.
Measure: Number; unit: participants
Arm/Group | Gufoni | Vibration | Sham
Number analyzed (Participants) | 70 | 67 | 72
participants | 51 | 46 | 38
Statistical Analysis 1: Comparison: Gufoni vs Sham; Test type: Superiority or Other; p = 0.02839, Regression, Logistic; Odds Ratio (OR) = 3.39, 95% CI 2-sided [1.58 to 7.31]
Statistical Analysis 2: Comparison: Vibration vs Sham; Test type: Superiority or Other; p = 0.0366, Regression, Logistic; Odds Ratio (OR) = 2.67, 95% CI 2-sided [1.25 to 5.67]

ADVERSE EVENTS:
Arm/Group | Gufoni | Vibration | Sham
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72 | 0/73
Other Adverse Events (participants affected / at risk) | 0/72 | 0/72 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No